CLINICAL TRIAL: NCT03914664
Title: Neural Correlates of Sensory Phenomena in Tourette Syndrome
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: NCoSPTS
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Tourette Syndrome; Sensory Disorders; Hypersensitivity; Tics
MeSH Terms: conditions — Tourette Syndrome; Sensation Disorders; Hypersensitivity; Tics | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tourette Syndrome: Adults (>18 years of age) with diagnosis of Tourette syndrome
  Interventions: Diagnostic Test: Electroencephalogram (EEG) testing procedure; Diagnostic Test: Autonomic function testing procedure
- Healthy Control: Adults who are generally healthy with no known neurologic or psychiatric diagnoses
  Interventions: Diagnostic Test: Electroencephalogram (EEG) testing procedure; Diagnostic Test: Autonomic function testing procedure

INTERVENTIONS:
Diagnostic Test: Electroencephalogram (EEG) testing procedure — EEG testing procedure, comprised of somatosensory and auditory event-related potential paradigms, as well as resting state EEG
Diagnostic Test: Autonomic function testing procedure — Autonomic function testing procedure, comprised of electrodes to determine heart rate variability and electrodermal activity (EDA)

SUMMARY:
The most pervasive sensory manifestation of TS is sensory over-responsivity (SOR). SOR is defined as excessive behavioral response to commonplace environmental stimuli. SOR is an integral but poorly understood facet of the TS phenotype, one intertwined with core elements of the disorder and worse QOL. This proposal seeks to clarify the mechanistic bases of SOR in TS. Adults with with TS will be recruited 1) to complete a standardized clinical symptom assessment battery and 2) to undergo electroencephalogram (EEG), autonomic, and audio-visual monitoring during tactile and auditory stimuli paradigms, as well as at rest.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a multifaceted disorder that affects 0.6-1% of the global population. Across the lifespan, individuals with TS suffer worse quality of life (QOL) than the general population. While tics are the defining feature of TS, it is the widespread psychiatric and sensory symptoms that exert greater impact on QOL: more than 85% of individuals with TS are diagnosed with a psychiatric disorder, and 90% experience distressing sensory symptoms. The latest TS disease models and practice guidelines account for common psychiatric symptoms, but sensory symptoms remain under-recognized and under-studied. Progress in understanding and treating TS requires deepening insight into the disorder's sensory dimension.

The most pervasive sensory manifestation of TS is sensory over-responsivity (SOR). SOR is defined as excessive behavioral response to commonplace environmental stimuli. SOR is associated with avoidant behavior and functional impairment. More than 50% of children and 80% of adults with TS report SOR. Across age groups, SOR is positively correlated with severity of tics and psychiatric symptoms and negatively correlated with QOL. Thus, SOR is an integral facet of the TS phenotype, one intertwined with core elements of the disorder and worse QOL. This proposal seeks to clarify the mechanistic bases of SOR in TS (Aims 1 and 2).

Enhanced understanding of SOR's neurobiological basis is crucial to a more complete knowledge of TS pathophysiology. Two neurophysiologic mechanisms are implicated in SOR: sensory gating impairment and autonomic hyperarousal. Sensory gating is the physiologic process whereby redundant environmental stimuli are filtered out in the early stages of perception. Impairment of sensory gating gives rise to altered sensory perception. Autonomic hyperarousal is a state of excessive sympathetic tone and/or reduced parasympathetic tone, which hampers behavioral adaptation to sensory input. In TS, multiple lines of evidence suggest both sensory gating and autonomic function are impaired. However, prior investigations have suffered from methodologic limitations and have not examined the link between neurophysiologic dysfunction and sensory symptoms.

Aim 1. Identify an electroencephalographic (EEG) signature of SOR in TS. Hypotheses: (1a) relative to healthy controls, TS adults exhibit impaired sensory gating; (1b) extent of impaired sensory gating in TS correlates with degree of SOR. We will recruit 60 TS adults and 60 age- and sex-matched healthy controls to complete rating scales for SOR, psychiatric symptoms, and tics. Subjects will then be monitored on dense-array scalp EEG during sequential auditory and tactile sensory gating paradigms.

Aim 2. Identify an autonomic signature of SOR in TS. Hypotheses: (2a) relative to healthy controls, TS adults exhibit autonomic hyperarousal in response to non-aversive sensory stimuli; (2b) extent of autonomic hyperarousal correlates with SOR severity in TS. Heart rate and electrodermal activity will be monitored during the Aim 1 sensory gating paradigms and during a 10-minute rest period. Heart rate variability and electrodermal activity will serve as indices of parasympathetic and sympathetic activity, respectively.

Impact: Results will clarify the extent of sensory gating impairment in TS, the nature of autonomic dysfunction in TS, and the clinical correlates of neurophysiologic dysfunction in TS.

ELIGIBILITY:
Inclusion criteria for TS arm:

* Diagnosis of Tourette syndrome or other chronic tic disorder
* ≥ 18 years of age
* Ability to complete survey instruments
* English fluency (given that all scales are validated in English)

Exclusion criteria for TS arm:

- Known diagnosis of autism spectrum disorder, developmental delay, cerebral palsy, other significant neurologic disease, schizophrenia, or psychotic disorders will be excluded, in order to lessen potentially confounding factors.

(Note: Patients with OCD, ADHD, anxiety, and/or depression will be permitted, given that these diagnoses are widely prevalent in the adult TS population.)

* Use of anti-seizure medications, stimulants, or other psychotropic medications known to alter EEG signal
* Recreational substance use within past 30 days

Inclusion criteria for healthy control arm:

* ≥ 18 years of age AND age within 5 years of a participant in the TS arm of same biological sex (for purposes of age- and sex-matching)
* Ability to complete survey instruments
* English fluency (given that all scales are validated in English)

Exclusion criteria for healthy control arm:

* Any neurologic or psychiatric diagnoses
* History of tics
* Use of any psychotropic medications within the past 30 days
* Recreational substance use within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The two groups of participants will include:
  1. adult with Tourette syndrome or other chronic tic disorder
  2. healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Network oscillations in response to sensory stimuli | Baseline
  Neural activity captured on EEG can be spectrally decomposed into various frequency constituencies. Neural activity in the gamma frequency range, so-called gamma band oscillations (GBOs), are associated with sensory processing and integration and are postulated to underlie sensory phenomena in TS.
Heart rate variability | Baseline
  Change beat-to-beat variability in heart rate
Electrodermal activity in response to sensory stimuli | Baseline
  Sweat response changes within 1-3 seconds of non-aversive sensory stimulus

SECONDARY OUTCOMES:
Premonitory Urge to Tic Scale (PUTS) | Within 1 week of baseline
  Validated self-report questionnaire comprised of 9 items assessing character and severity of premonitory urges. Scale range: 9 (least affected) - 36 (most affected)
Yale Global Tic Severity Scale (YGTSS) | Within 1 week of baseline
  Validated, gold-standard clinician-administered tic assessment scale, comprised of 11 items. Scale range: 0 (best) - 100 (worst)
Dimensional Obsessive Compulsive Scale (DOCS) | Within 1 week of baseline
  Validated self-report questionnaire assessing severity of obsessive and compulsive symptoms, comprised of 20 items. Scale range 0 (least affected) - 80 (most affected)
Adult ADHD Self-Report Screening Scale | Within 1 week of baseline
  Validated self-report scale, developed since release of Diagnostic and Statistical Manual-V, comprised of 6 items. Scale range 0 (least affected) - 24 (most affected)
Generalized Anxiety Disorder 7 (GAD-7) | Within 1 week of baseline
  Validated self-report scale assessing presence and extent of anxiety, comprised of 7 items. Scale range 0 (least affected) - 21 (most affected)
Patient Health Questionnaire 9 (PHQ-9) | Within 1 week of baseline
  Validated self-report scale assessing presence and extent of depression, comprised of 9 items. Scale range 0 (least affected) - 27 (most affected)
Sensory Gating Inventory (SGI) | Within 1 week of baseline
  Validated self-report questionnaire assessing sensory hypo- or hyper-sensitivity, comprised of 36 items. The 4 sub-scales include Perceptual Modulation, Distractability, Over-Inclusion, and Fatigue and Stress Vulnerability. Total scale range 0 (least affected) - 180 (most affected)
Sensory Perception Quotient (SPQ) | Within 1 week of baseline
  Validated self-report questionnaire assessing sensory hypo- or hyper-sensitivity, comprised of 35 items. Scale range 0 (highest sensory sensitivity) - 105 (lowest sensory sensitivity).
Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL) | Within 1 week of baseline
  Validated self-report questionnaire assessing health-related quality of life for patients with Tourette syndrome, comprised of 27 items. Scale range 0 (best quality of life) - 108 (worst quality of life)
Patient Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment | Within 1 week of baseline
  Validated self-report questionnaire to measures sleep-related impairments, consisting of 8 items. Scale range 0 - 100 (t-score scaled with lower values indicating less impairment).
Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) | Within 1 week of baseline
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 37 items. Each scale item is a statement to which respondents must select "never" (0) to "always" (5) on a six-point Likert scale. No total MAIA-2 score exists. Rather, individual scale items belong to one of eight MAIA-2 subscales. For each subscale, higher score signifies more of that construct.
Body Perception Questionnaire - Short Form (BPQ-SF) | Within 1 week of baseline
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 46 items total, divided into 3 sections: Body Awareness (raw total score 26-130), Supradiaphragmatic Reactivity (raw total score 15-69), and Subdiaphragmatic Reactivity (raw total score 6-28). Raw scores are converted to T-scores. Higher raw and T-scores indicate greater maladaptive body awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical variables, EEG data, and autonomic data metrics may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The above information will be available for sharing within 6 months of publication.
Access Criteria: Researchers wishing to access the above information should contact the investigative team and provide: 1) hypothesis-driven scientific question for which the data will be analyzed and 2) proposed methods for responsibly analyzing the data.